CLINICAL TRIAL: NCT06533540
Title: A Single-center, Single Group, Dose Escalation, Phase 1 Clinical Trial to Investigate the Safety of TPX-121 in Subjects With Moderate-to-Extreme Nasolabial Folds
Brief Title: Safety Study of TPX-121 on Nasolabial Folds
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-TPX-121-23-01
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Nasolabial Fold, Hypoplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low dose (Experimental)
  Interventions: Biological: TPX-115(allogeneic fibroblasts)
- middle dose (Experimental)
  Interventions: Biological: TPX-115(allogeneic fibroblasts)
- high dose (Experimental)
  Interventions: Biological: TPX-115(allogeneic fibroblasts)

INTERVENTIONS:
Biological: TPX-115(allogeneic fibroblasts) — Intradermal injection of TPX-115(allogeneic fibroblasts)

SUMMARY:
Nasolabial folds augmentation is possible through dermal filler and botulinum toxin, however, safety issues are existed as well as efficacy. Therefore, there is a need for a safer procedure for nasolabial folds correction. This study (Project No. TPX-121) assesses the safety of allogeneic fibroblasts (TPX-115) on nasolabial folds. The safety endpoint is dose-limiting toxicity (DLT). In addition, exploratory endpoints are the improvement of nasolabial folds in Wrinkle Severity Rating Scale (WSRS) at week 4 and 12, change in WSRS and Wrinkle Severity Scale (WSS) at week 4 and 12, and overall appearance improvement rate in Global Aesthetic Improvement Scale (GAIS) at week 4 and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Be 19 years old or older
2. Have confirmed nasolabial folds severity equal to or more than grade 3 evaluated by WSRS and WSS at face to face evaluation.
3. Have unsatisfied or very unsatisfied nasolabial folds.
4. Voluntarily sign the informed consent for participation in the study.

Exclusion Criteria:

Current disease and medical history

1. Inflammatory and infectious skin diseases, unhealed wounds and scars (e.g. Keloids), or benign tumor on nasolabial folds.
2. Chronic skin diseases (e.g. Psoriasis, Atopic dermatitis).
3. Genetic diseases that affect fibroblasts or collagen (e.g. Achondroplasia, Osteogenesis imperfecta).
4. Autoimmune diseases.
5. Active hepatitis B or C (However, in the case of simple carriers or hepatitis B, except when the antiviral agent was stably taken for 6 months prior to screening).
6. Human immunodeficiency virus (HIV) positive.
7. Coagulopathy.
8. History of malignant tumors within the last 5 years.
9. Anaphylaxis or severe combined allergy
10. Have allergies to bovine proteins or gentamicin.
11. Acute or chronic infectious diseases.
12. Severe heart diseases (e.g. Myocardial infarction, Heart failure), severe liver diseases (e.g. Cirrhosis, Liver failure), or severe renal diseases (e.g. Kidney failure).
13. Hypersensitivity to amide-based local anesthetics (However, those who agree not to use local anesthetics can register).

    Prohibited drugs and treatments.
14. Administered systemic corticosteroids within 12 weeks prior to screening or is scheduled to be administered for at least 2 weeks during the study.
15. Treated cell therapy or stem cell therapy within 1 year prior to screening.
16. Surgical procedures or surgeries such as fillers or fat grafting on facial part within 1 year prior to screening.
17. Surgical procedures or surgeries of permanent fillers on facial part prior to screening.
18. Surgical procedures or surgeries of botulinum toxin injection or face lift surgery on facial part within 6 months prior to screening.
19. Planned facial cosmetic surgery to improve nasolabial folds during the study.

    Laboratory inspection
20. Those who fall under the following figures during screening. 1) White blood cell < 4.5x10^3/ul and > 11.0x10^3/ul 2) Platelet count < 100,000/mm^3 3) Hemoglobin < 9g/dL

    Other
21. Disagree to take pictures of nasolabial folds
22. Be pregnant, breastfeeding, planning pregnancy or unwilling to use of contraceptice.
23. Have participated in other clinical trials and recevied investigational products/devices within 30 days of this study.
24. Be deemed inadequate for the study by investigators(e.g. A person with severe asymmetry in the lower echocardiogram).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Week 4
  The number of subjects evaluated grade 3 or higher adverse drug reactions according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0

OTHER OUTCOMES:
Improvement WSRS grade from baseline | Week 4 and Week 12
  Improvement Wrinkle Severity Rating Scale (WSRS) grade of nasolabial folds from baseline evaluated by an investigator based on pictures taken at week 4 and 12.
  The WSRS ranges from 1 (absent) to 5 (Extreme). A negative change from baseline indicates improvement.
WSRS grade change from baseline | Week 4 and Week 12
  Wrinkle Severity Rating Scale (WSRS) grade change from baseline evaluated by an investigator based on pictures taken at week 4 and 12.
  The WSRS ranges from 1 (absent) to 5 (Extreme). A negative change from baseline indicates improvement.
WSS grade change from baseline | Week 4 and Week 12
  Wrinkle Severity Scale (WSS) grade change from baseline evaluated by an investigator based on pictures taken at week 4 and 12.
  The WSS ranges from 0 (absent) to 5 (Extreme). A negative change from baseline indicates improvement.
Overall appearance improvement percentage(%) using GAIS | Week 4 and Week 12
  Overall appearance improvement percentage(%) rated by subjects using Global Aesthetic Improvement Scale (GAIS) at week 4 and 12.
  In the case of overall appearance improvement rate using GAIS being +3 point (Very much improved), +2 (Much improved), or +1 (Improved)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyun Chung, M.D., Principal Investigator — Kyungpook National University, School of Medicine
Locations (1):
- Kyungpook National University, School of Medicine, Daegu, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No